CLINICAL TRIAL: NCT02614495
Title: A Multi-center , Opened, Phase II Study of Safety and Efficacy of Sulfatinib in Advanced Medullary Thyroid Carcinoma ( MTC) and Iodine-refractory Differentiated Thyroid Carcinoma (DTC)
Brief Title: Study of Sulfatinib in Treating Advanced Medullary Thyroid Carcinoma and Iodine-refractory Differentiated Thyroid Carcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hutchison Medipharma Limited (Industry)
Responsible Party: Sponsor
Organization: Hutchmed (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2015-012-00CH2
Record Dates: First submitted 2015-11-24; First posted 2015-11-25 (Estimated); Last update posted 2020-02-13 (Actual); Status verified 2019-11

CONDITIONS: Thyroid Carcinoma
MeSH Terms: conditions — Thyroid Neoplasms | interventions — surufatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Surufatinib (Experimental): 300mg once-daily
  Interventions: Drug: Surufatinib

INTERVENTIONS:
Drug: Surufatinib — Patients receive oral Sulfatinib at a dose of 300mg/d within 1 hour after breakfast (once-daily dosing continuously, every 28-day treatment cycle)
  Other Names: HMPL-012; Sulfatinib

SUMMARY:
A multi-center , opened, Phase II study to assess the efficacy and safety of Sulfatinib 300 mg Sulfatinib in advanced Medullary Thyroid Carcinoma ( MTC) and iodine-refractory differentiated thyroid carcinoma (DTC).

DETAILED DESCRIPTION:
This study adopt Simon's two-stage designs method. In the first stage, When the first 12 patients enrolled complete therapy of Cycle 1, investigators and sponsors will analyze safety and pharmacokinetic (PK) data, to determine whether the dose is suitable for TC and enrollment should be stopped during this period.15 subjects will be enrolled in both subgroups (advanced MTC and iodine-refractory DTC), and more 10 subjects in each subgroups will be enrolled after efficacy assessment in the second stage.

Patients receive oral sulfatinib at a dose of 300mg/d within 1 hour after breakfast (once-daily dosing continuously, every 28-day treatment cycle) until disease progression, death, or intolerable toxicity, or in the opinion of the investigator, patients were no longer deriving clinical beneﬁt、lost to follow-up、withdrew informed consent form, or sponsors terminated the study, whichever comes first.

ELIGIBILITY:
Inclusion Criteria:

1. Informed consent must be obtained in writing for all subjects before enrollment into the study;
2. Age 18 years or older
3. Subjects must have histologically or cytologically confirmed diagnosis of locally advanced and/ or metastatic MTC or iodine-refractory DTC (papillary, follicular , Hürthle cell and other variable type carcinoma), losing the surgical indications or can't undertake external radiotherapy
4. Subjects must show evidence of disease progression within 12 months (assessed and confirmed by central radiographic review of CT and/or MRI scans) before initial treatment of this study
5. Subjects must be I-refractory / resistant as defined by at least one of the following: One or more measurable lesions that has progressed by CT and/or MRI scans within 12 months of Iodine-131 (131I) therapy; One or more measurable lesions that do not demonstrate 131I uptake on any radioiodine scan ; Cumulative activity of 131I of > 600 millicurie or 22 gigabecquerel (GBS), and independently reviewed radiologic evidence of progression within the previous 12 months before initial treatment of this study
6. At least 6 months of last dose administered prior to study treatment
7. Subjects may have received 0 or 1 prior vascular endothelial growth factor (VEGF)/VEGFR-targeted therapy (for example , patients with MTC have received vandetanib or cabozantinib; patients with DTC have received sorafenib or lenvatinib) or other targeted inhibitors
8. Subjects with DTC, serum thyroid-stimulating hormone (TSH) concentration should be lower than 0.1 milliunits per litre (mU/L) (or other corresponding units) before enrollment into the study; Subjects with MTC, levels of serum TSH concentration should be in the normal range
9. Subjects must have an Eastern Cooperative Oncology Group (ECOG) Performance Status of 0-1
10. Subjects must have measurable lesions meeting the criteria of Response Evaluation Criteria in Solid Tumors (RECIST) 1.1
11. The expecting life scan was more than 12 weeks
12. Females or Males of childbearing potential must agree to use a highly effective method of contraception (e.g., a double-barrier method, condom, a injective or oral contraceptive, an intrauterine device) throughout the entire study period and for 90 days after study drug discontinuation. All females will be considered to be of childbearing potential unless they are postmenopausal.

Exclusion Criteria:

1. Absolute neutrophil count 1.5×109/L, or platelet<100 ×109/L, or hemoglobin< 9g/dL
2. Serum bilirubin >1.5 the upper limit of normal (ULN)
3. Serum alanine transaminase (ALT) , aspartate aminotransferase (AST) or Alkaline phosphatase (ALP) ≥2.5 ULN (Patients with documented disease infiltration of the liver may have ALT, AST or ALP levels ≥ 5 the ULN)
4. Serum creatinine≥1.5 the upper limit of normal (ULN) , or estimated creatinine clearance < 60 mL/min
5. Subjects having≥2+ proteinuria on urine dipstick testing will undergo 24h urine collection for quantitative assessment of proteinuria. Subjects with urine protein≥1g/24 h will be ineligible
6. International normalized ratio (INR) ≥1.5 the ULN or activated partial thromboplastin time (aPTT) ≥1.5 the ULN (For patients requiring anticoagulation therapy with warfarin, a stable INR between 2-3 is required)
7. Serum potassium, calcium (albumin-bound ionic or corrected) or magnesium exceed the normal range with clinical significance
8. Active hypertension (systolic pressure≥140mm Hg, or diastolic pressure ≥90mm Hg) that drugs can't control
9. Gastrointestinal disease or condition that investigators suspect may affect drug absorption, including but not limited to, previously subtotal gastrectomy surgery, active gastric and duodenal ulcers, ulcerative colitis and other digestive disease, gastrointestinal tumor with active bleeding, or other gastrointestinal conditions that may cause bleeding or perforation by investigator's discretion
10. History or presence of a serious hemorrhage (>30 ml within 3 months), hemoptysis (>5 ml blood within 4 weeks) or a thromboembolic event (including transient ischemic attack) within 12 months
11. Clinically significant cardiovascular disease, including but not limited to, acute myocardial infarction within 6 months prior to enrollment, severe/unstable angina pectoris or coronary artery bypass grafting, congestive heart failure according to the New York Heart Association (NYHA) classification ≥ 2; ventricular arrhythmias which needs drug treatment; LVEF (LVEF) <50%
12. Prolongation of QT interval to≥480 ms
13. Active malignancy (except for definitively treated melanoma in-situ, basal or squamous cell carcinoma of the skin, or carcinoma in-situ of the cervix) within the past 5 years
14. Patients were excluded from the study if they had received anti-tumor therapies, including but not related to chemotherapy, radial radiation therapy, biological therapy, immunotherapy, or treatment with herb product within 4 weeks prior to initial treatment of this study. TSH suppression therapy is not included
15. Patients receive palliative irradiation for the bone metastasis within 2 weeks prior to before initial treatment of this study
16. Patients receive cytochrome P450 3A4 (CYP3A4) strong inducer or inhibitors (as seen in attachment 3) within 2 weeks (3 weeks for Hypericum perforatum) prior to initial treatment of this study
17. Clinically significant and active infection, including but not limited to HIV infection
18. Clinically significant history of liver disease, including virus hepatitis [known HBV carrier, active hepatitis B virus (HBV) infection (>1*104/ml) must be excluded; known hepatitis C virus (HCV) carrier, active HCV infection (>1*103/ml) must be excluded] and other hepatitis, cirrhosis
19. Major surgery within 4 weeks prior to enrollment, or the incision is still not fully healed
20. Subjects with known brain metastases or spinal cord compression who have not completed radiosurgery or surgical resection, or who have previously treated but with no clinical imaging evidence of disease stability
21. Subjects has not recovered from any toxicity related to previous anticancer treatment to level 0 or 1 (alopecia excluded)
22. Subjects who have received any investigational agent within 4 weeks prior to the first dose of study drug
23. Pregnancy (test is positive before the first dose of study drug) or any other lactating women
24. Any other diseases, metabolic dysfunction, physical examination finding, or clinical laboratory finding that, in the investigator's opinion, gives reasonable suspicion of a disease or condition that contraindicates the use of an investigational drug or that may affect the interpretation of the results or renders the patient at high risk from treatment complications.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2016-02-24 (Actual); Primary Completion 2018-09-30 (Actual); Study Completion 2018-09-30 (Actual)

PRIMARY OUTCOMES:
objective response rate (ORR) | 16 months after the last patient enrolled
  the incidence of confirmed complete response or partial response

SECONDARY OUTCOMES:
Adverse events evaluated by the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) v4.03 | From first dose to within 30 days after the last dose
  The safety and tolerability of sulfatinib will be evaluated based on adverse events data. Other safety parameters include physical examination, vital signs, laboratory test results (i.e., hematology, chemistry panel, and urinalysis), 12-lead electrocardiogram, and ultrasonic cardiogram
The disease control rate (DCR) | 16 months after the last patient enrolled
  the incidence of complete response, partial response and stable disease
Progression Free Survival (PFS) | 16 months after the last patient enrolled
  the duration between the randomization date and the first disease progression (PD) or death (whichever comes first).
Time to Response (TTR) | 16 months after the last patient enrolled
  the period from the date of randomization to the date when the criteria for complete response or partial response was first measured (first record shall prevail).

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Peking Union Medical College Hospital, Beijing, Beijing Municipality
  - Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality